CLINICAL TRIAL: NCT01044069
Title: A Phase I Trial of Precursor B Cell Acute Lymphoblastic Leukemia (B-ALL) Treated With Autologous T Cells Genetically Targeted to the B Cell Specific Antigen CD19
Brief Title: Precursor B Cell Acute Lymphoblastic Leukemia (B-ALL) Treated With Autologous T Cells Genetically Targeted to the B Cell Specific Antigen CD19
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-114
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia
Keywords: Cyclophosphamide; T cell; leukapheresis; stem cell transplant; bone marrow transplant; 09-114
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pts with B Cell Acute Lymphoblastic Leukemia (Experimental): This is a phase I study. Patients with CD19+ ALL (CR, relapsed, MRD, or refractory) are eligible for enrollment. B-ALL patients in first CR will be enrolled but only treated if they develop MRD or a frank relapse, while patients with MRD or with documented relapsed/refractory disease are eligible for immediate treatment. The T cell doses originally proposed in this study were based on doses administered safely in prior autologous T cell adoptive therapy trials but the dose has been modified based on the toxicities observed in patients with morphologic evidence of disease. Patients will be treated with different doses of T cells depending on the amount of disease at the time of T cell infusion. Patients in Cohort 1 (<5% blasts in the BM) will continue to receive 10^6 19-28z+ T cells/kg as previously. Patients in Cohort 2 (≥5% blasts in the BM) will receive the reduced dose of 1x106 19-28z+ T cells/kg).
  Interventions: Biological: gene-modified T cells targeted

INTERVENTIONS:
Biological: gene-modified T cells targeted — Pts will undergo leukapheresis. The leukapheresis product will be washed & frozen until the GTF is directed to start T cell production by the PI. CD3+ T cells will be isolated from the leukapheresis, & transduced with the 19-28z chimeric receptor & expanded. All relapsed (either MRD+ or morphologic) & refractory pts get re-induction chemo whenever feasible to optimally reduce the tumor burden prior to the T cell infusion. The re-induction chemo regimen will be selected by the treating dr. based on prior therapy, adverse reactions to chemo & highest likelihood to achieve an optimal response. Once pts recover from the toxicities of the re-induction chemo the disease status will be re-evaluated by repeating bone marrow aspirate or biopsy. Pts get conditioning chemo (min 2 weeks from end of re-induction chemo) followed 2-7 days later by the 19-28z+ T cells. Pts will be tx in 2 cohorts with diff doses of T cells according to the amount of disease immediately prior to the T cell infusion.

SUMMARY:
This study is an investigational approach that uses immune cells, called "T cells", to kill leukemia. These T cells are removed from blood, modified in a laboratory, and then put back in the body. T cells fight infections and can also kill cancer cells in some cases. However, right now T cells are unable to kill the cancer cells. For this reason we will put one gene into the T cells that allows them to recognize and kill the leukemia cells. This gene will be put in the T cells by a weakened virus. The gene will produce proteins in the T cells that help the T cells recognize the leukemia cells and possibly kill them. The doctors have found that T cells modified in this way can cure an ALL-like cancer in mice.

The main goals of this study is to determine the safety and appropriate dose of these modified T cells in patients with ALL. This will be done in a "clinical trial." The dose of modified T-cells will depend on if you have disease present in your bone marrow or not. The patient will also receive chemotherapy before the T cells. We will use normally chemotherapy that is used in patients with leukemia. The chemotherapy is given to reduce leukemia and to allow the T cells to live longer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients are eligible (> or = to 18 year old).
* Patients must have B- ALL refractory, relapsed, MRD, or in first CR as described below.
* Complete remission is defined as restoration of normal hematopoiesis with a neutrophil count > 1,000 x 106/L, a platelet count > 100,000 x 106/L, and hemoglobin > 10 g/dL. Blasts should be < 5% in a post-treatment bone marrow differential. Furthermore, there should be no clinical evidence of leukemia for a minimum of four weeks.
* MRD is defined as patients meeting the criteria for CR above, but with residual disease measured by a quantitative PCR, or by flow or by deep-sequencing of the IgH rearrangements . The assay from blood and/or bone marrow defines MRD by qPCR as a cycle threshold (CT) that is at least 1 CT value < than the lowest CT value from the background. Outside laboratory tests may suffice for this assessment at the discretion of the Principal Investigator.

Relapsed B-ALL will be defined as patients that meet the above criteria for a CR before developing recurrent disease (increased bone marrow blasts). Refractory patients will be defined as patients that have not achieved a CR after 1 cycle of induction chemotherapy

* Patients must have a diagnosis of B-ALL by flow cytometry, or bone marrow histology, and/or cytogenetics.
* Patients must have CD19+ ALL as confirmed by flow cytometry and/or immunohistochemistry.
* Creatinine < 2.0 mg/100 ml, bilirubin < 2.0 mg/100 ml, AST and ALT < 3x normal, PT and PTT < 2x normal outside the setting of stable chronic anticoagulation therapy. LFTs (Bilirubin, AST, and/or ALT) may be acceptable if the elevation is secondary to leukemia infiltration or leukemia therapy with tyrosine kinase inhibitors.
* Adequate cardiac function (LVEF ≥ 40%) as assessed by ECHO or MUGA or other similar cardiac imaging performed within 1 month of enrollment.
* Adequate pulmonary function as assessed by ≥ 92% oxygen saturation on room air by pulse oximetry.
* Patients must have adequate access for leukapheresis procedure as assessed by staff from the MSKCC Donor Room.
* Life expectancy > 3 months

Exclusion Criteria:

* Karnofsky performance status < 70.
* Active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF) or symptomatic CNS leukemia (i.e. cranial nerve palsies or other significant neurologic dysfunction) within 28 days of enrollment. Prophylactic intrathecal medication is not a reason for exclusion.
* Patients previously treated with an allogeneic SCT that is currently complicated by active GVHD requiring T cell suppressive therapy.

Patients with following cardiac conditions will be excluded:

* New York Heart Association (NYHA) stage III or IV congestive heart failure
* Myocardial infarction ≤6 months prior to enrollment
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* History of severe non-ischemic cardiomyopathy with EF ≤20%

  * Patients with HIV, hepatitis B or hepatitis C infection.
  * Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2010-01-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of adoptive transfer of gene-modified autologous CD19-specific T cells in adult patients with B-ALL. | 2 years

SECONDARY OUTCOMES:
To assess the anti-leukemic effect of adoptively transferred anti-CD19 T cells. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Valtis YK, Lin C, Nemirovsky D, Devlin SM, Rejeski K, Curran KJ, Wang X, Shah NN, Jeyakumar N, Miller K, Zhang A, Kota VK, Al Darobi A, Muhsen IN, Sasine JP, Aldoss I, Advani AS, Reshef R, Chen EC, Kopmar NE, Tsai SB, Hilal T, Shah BD, Faramand RG, Solh MM, Tan V, Bezerra ED, Battiwalla M, Ramakrishnan A, Mathews J, Shaughnessy PJ, Mountjoy L, Hoeg RT, Dykes KC, Logan AC, Kumaran M, Schwartz MS, Tracy SI, Moore J, Odstrcil Bobillo S, Frey NV, Connor MP, Ladha A, Dholaria B, Sutherland KC, Roloff GW, Muffly LS, Park JH. CAR HEMATOTOX independently predicts outcomes after CD19 CAR-T therapy for acute lymphoblastic leukemia. Blood Adv. 2025 Oct 6:bloodadvances.2025017526. doi: 10.1182/bloodadvances.2025017526. Online ahead of print. PMID 41052404
- [Derived] Jain T, Knezevic A, Pennisi M, Chen Y, Ruiz JD, Purdon TJ, Devlin SM, Smith M, Shah GL, Halton E, Diamonte C, Scordo M, Sauter CS, Mead E, Santomasso BD, Palomba ML, Batlevi CW, Maloy MA, Giralt S, Smith E, Brentjens R, Park JH, Perales MA, Mailankody S. Hematopoietic recovery in patients receiving chimeric antigen receptor T-cell therapy for hematologic malignancies. Blood Adv. 2020 Aug 11;4(15):3776-3787. doi: 10.1182/bloodadvances.2020002509. PMID 32780846
- [Derived] Pennisi M, Jain T, Santomasso BD, Mead E, Wudhikarn K, Silverberg ML, Batlevi Y, Shouval R, Devlin SM, Batlevi C, Brentjens RJ, Dahi PB, Diamonte C, Giralt S, Halton EF, Maloy M, Palomba ML, Sanchez-Escamilla M, Sauter CS, Scordo M, Shah G, Park JH, Perales MA. Comparing CAR T-cell toxicity grading systems: application of the ASTCT grading system and implications for management. Blood Adv. 2020 Feb 25;4(4):676-686. doi: 10.1182/bloodadvances.2019000952. PMID 32084260
- [Derived] Park JH, Romero FA, Taur Y, Sadelain M, Brentjens RJ, Hohl TM, Seo SK. Cytokine Release Syndrome Grade as a Predictive Marker for Infections in Patients With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia Treated With Chimeric Antigen Receptor T Cells. Clin Infect Dis. 2018 Aug 1;67(4):533-540. doi: 10.1093/cid/ciy152. PMID 29481659
- [Derived] Park JH, Riviere I, Gonen M, Wang X, Senechal B, Curran KJ, Sauter C, Wang Y, Santomasso B, Mead E, Roshal M, Maslak P, Davila M, Brentjens RJ, Sadelain M. Long-Term Follow-up of CD19 CAR Therapy in Acute Lymphoblastic Leukemia. N Engl J Med. 2018 Feb 1;378(5):449-459. doi: 10.1056/NEJMoa1709919. PMID 29385376
- [Derived] Brentjens RJ, Riviere I, Park JH, Davila ML, Wang X, Stefanski J, Taylor C, Yeh R, Bartido S, Borquez-Ojeda O, Olszewska M, Bernal Y, Pegram H, Przybylowski M, Hollyman D, Usachenko Y, Pirraglia D, Hosey J, Santos E, Halton E, Maslak P, Scheinberg D, Jurcic J, Heaney M, Heller G, Frattini M, Sadelain M. Safety and persistence of adoptively transferred autologous CD19-targeted T cells in patients with relapsed or chemotherapy refractory B-cell leukemias. Blood. 2011 Nov 3;118(18):4817-28. doi: 10.1182/blood-2011-04-348540. Epub 2011 Aug 17. PMID 21849486
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm